CLINICAL TRIAL: NCT06792916
Title: Evaluation of Subgingival Mechanical Periodontal Therapy with the Additional Local Application of a Spermidine-Based Gel
Brief Title: This Study Evaluates the Clinical Effect of Adding Spermidine Gel to Minimally Invasive Non-surgical Periodontal Therapy (MINST) to Improve Periodontal Health.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Luca Ramaglia (Other)
Responsible Party: Sponsor-Investigator, Luca Ramaglia, Professor, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 342/2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Peridontitis
MeSH Terms: interventions — Spermidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MINST plus spermidine gel (Experimental)
  Interventions: Procedure: spermidine and minimally invasive non surgical tecnique
- MINST (minimally invasive non surgical tecnique) (Active Comparator)
  Interventions: Other: peridontal therapy (minimally invasive non surgical tecnique)

INTERVENTIONS:
Procedure: spermidine and minimally invasive non surgical tecnique — minimally non surgical periodontal therapy will be performed with the adjunct of spermidine based gel
  Arms: MINST plus spermidine gel
Other: peridontal therapy (minimally invasive non surgical tecnique) — subgingival instrumentation will be performed according to MINST
  Arms: MINST (minimally invasive non surgical tecnique)

SUMMARY:
This study investigates the effectiveness of using a spermidine-based gel as an adjunct to minimally invasive non-surgical periodontal therapy (MINST) for treating periodontitis. The primary outcome is to assess whether the addition of spermidine gel reduces pocket depth (PPD) compared to MINST alone. Secondary outcome include evaluating other periodontal parameters like bleeding on probing, FMBS and FMPS and CAL over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older. Presence of untreated periodontitis with at least 2 sites showing clinical attachment loss (CAL) > 2 mm and probing depth (PD) > 4 mm.

Voluntary signing of informed consent.

Exclusion Criteria:

Presence of systemic diseases (e.g., diabetes mellitus, cardiovascular, renal, hepatic, or pulmonary conditions).

Smokers (≥10 cigarettes per day). Pregnancy or breastfeeding. Allergy to any ingredients in the products used in the study. Diseases affecting bone and/or connective tissue metabolism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Probing depth (PD) | From non surgical periodontal therapy to 6 months
  peridontal probing depth

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Federico II, Naples, Italy, Italy